CLINICAL TRIAL: NCT01914367
Title: Study of the Molecular Mechanisms Underlying the Cross-neutralizing Capacity of AS04-adjuvanted HPV Vaccine (Cervarix®) in Comparison With the Aluminiumhydroxyphosphate Sulphate Adjuvanted HPV Vaccine (Gardasil®)
Acronym: HPVXneutra001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013/422; 2013-002340-90 (EudraCT Number)
Record Dates: First submitted 2013-06-06; First posted 2013-08-02 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Infection With Human Papillomavirus
MeSH Terms: interventions — human papillomavirus vaccine, L1 type 16, 18; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervarix group (Active Comparator): One sib of each twin pair will be given Cervarix according to the 0, 1, 6 month vaccination scheme.
  Interventions: Biological: cervarix
- Gardasil Group (Active Comparator): One sib of each twin pair will be given Gardasil according to the 0, 1, 6 month vaccination scheme.
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: cervarix — 3 doses will be given, one on Day 0, one on Day 30 and one on Day 180 ± 7 days, intramuscular in the deltoid muscle of the non-dominant arm
  Other Names: GSK's commercially available bivalent HPV types 16 and 18 recombinant vaccine containing AS04 adjuvant (Cervarix®)
  Arms: Cervarix group
Biological: Gardasil — 3 doses will be given, one on Day 0, one on Day 60 ± 2 days and one on Day 180 ± 7 days, intramuscular in the deltoid muscle of the non-dominant arm
  Other Names: Merck's commercially availably quadrivalent HPV(types 6, 11, 16, 18) recombinant vaccine containing amorphous aluminiumhydroxyphosphate sulphate adjuvant
  Arms: Gardasil Group

SUMMARY:
Six identical female twins aged 9-13 years will participate. One sib of each twin pair will be given Cervarix according to the 0, 1, 6 month vaccination scheme, while the other sib will be given Gardasil according to the 0, 2, 6 month vaccination scheme. Three blood samples will be taken (the first prior to vaccine administration, the second and third 7 days after dose 2 and 3, respectively). The blood samples will be used to determine: 1) the magnitude the anti-HPV 16 and anti-HPV-18 antibody responses, 2) as well as the cross-reactive pattern of these responses towards related, non-vaccine HPV strains (HPV-31 and -33, and HPV-45). 3) plasmablast isolated from blood taken 7 days after the 3rd dose in the first place (and eventually after the 2nd dose also) will be examined for for the usage of VDJ and VJ segments in the immunoglobulin heavy (VH) and light (VL) heavy and light chains. Gene useg in B cells induced by Cervarix and Gardasil will be compared. Finally the cross-reactive potential of monoclonal antibodies obtained by eukaryotic expression of a series of heavy (VH) and light (VL) chains from single ASC isolated after the 3rd dose of a three-dose schedule of either Cervarix or Gardasil will be examined.

The duration of the study is approximately 187 days. Five study visits will take place, over a time period of 6.5 months, followed by a telephone call after 12 months.

The purpose of the study is to learn more about the molecular mechanisms underlying the cross-neutralizing capacity of AS04-adjuvanted HPV vaccine (Cervarix®) in comparison with the aluminiumhydroxyphosphate sulphate adjuvanted HPV vaccine (Gardasil®).

ELIGIBILITY:
Inclusion Criteria:

* Six homozygous twins in good health, without preceding sexual activity (virgin). Subjects have a negative pregnancy test on the day of vaccination and have agreed to continue abstinence during the entire study period and for two months after completion of the vaccination series.

Exclusion Criteria:

* Subjects are not participating in any other clinical trials and have not been vaccinated previously against HPV and have not had an administration of MPL or AS04 in the past.

Ages: 9 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2015-09-23 (Actual)

PRIMARY OUTCOMES:
comparing of VDJ and VJ segments in the immunoglobulin heavy and light chains/plasmablasts | at day 187
comparing the mutational diversity that occurs following vaccine-induced affinity maturation in plasmablasts | at day 187

SECONDARY OUTCOMES:
evaluation of the cross-reactive pattern of polyclonal serum antibodies | at day 187
comparing of VDJ and VJ segment usage and affinity maturation in HPV-specific antibodies | at day 187
comparing of the cross-reactive potential of monoclonal antibodies obtained by eukaryotic expression of a series of heavy (VH) and light (VL) chains from single ASC | at day 187

CONTACTS AND LOCATIONS:
Overall Officials: Geert Leroux-Roels, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium